CLINICAL TRIAL: NCT04185948
Title: A Pilot Study Investigating the Acceptability and Impact of the Mediterranean Diet and Intermittent Fasting
Brief Title: Pilot Study on the Impact of the Mediterranean Diet and Intermittent Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Jose Lara Gallegos, Senior Lecturer, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLS-JLG-2019
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet plus intermittent fasting (Experimental): For 4 weeks participants will be encouraged to adopt the Mediterranean dietary guidelines as recommended by the Mediterranean Diet Foundation in Barcelona, Spain. In combination with these guidelines, an intermittent fasting regime involving two days of the week will be implemented. The regime will encourage individuals to consume of 500kcal per day for women and 625kcal per day for men, resulting in 75% daily caloric restriction during each of these two days.
  Interventions: Behavioral: Mediterranean diet guidelines plus intermittent fasting
- Eatwell guide plus intermittent fasting (Active Comparator): For 4 weeks participants will be encouraged to adopt the UK dietary guidelines (Eatwell Guide). In combination with these guidelines, an intermittent fasting regime involving two days of the week will be implemented. The regime will encourage individuals to consume of 500kcal per day for women and 625kcal per day for men, resulting in 75% daily caloric restriction during each of these two days.
  Interventions: Behavioral: UK Eatwell guidelines plus intermittent fasting

INTERVENTIONS:
Behavioral: Mediterranean diet guidelines plus intermittent fasting — For 4 weeks participants will be encouraged to adopt the Mediterranean dietary guidelines as recommended by the Mediterranean Diet Foundation in Barcelona, Spain. In combination with these guidelines, an intermittent fasting regime involving two days of the week will be implemented. The regime will encourage individuals to consume of 500kcal per day for women and 625kcal per day for men, resulting in 75% daily caloric restriction during each of these two days.
  Arms: Mediterranean diet plus intermittent fasting
Behavioral: UK Eatwell guidelines plus intermittent fasting — For 4 weeks participants will be encouraged to adopt the UK dietary guidelines (Eatwell Guide). In combination with these guidelines, an intermittent fasting regime involving two days of the week will be implemented. The regime will encourage individuals to consume of 500kcal per day for women and 625kcal per day for men, resulting in 75% daily caloric restriction during each of these two days.
  Arms: Eatwell guide plus intermittent fasting

SUMMARY:
This clinical trial attempts to evaluate the feasibility and acceptability of an intervention combining intermittent fasting and the Mediterranean diet guidelines vs an comparative intervention combining intermittent fasting but using the UK dietary guidelines.

Participants will be randomised to these intervention using a parallel design. Weight change and blood lipids will be assessed.

DETAILED DESCRIPTION:
This study will have a randomised parallel study comparing two interventions involving intermittent fasting. One of the interventions will use the Mediterranean dietary guidelines proposed by the Mediterranean Diet Foundation, the other intervention will use the UK dietary guidelines (Eatwell Guide).

In this study, the interventions will require participants to adopt these interventions for 4 weeks. A basic website containing support information will be develop for each of these interventions.

Baseline measurements will be taken at the start of the study. Blood samples will be obtained in a fasted state before and after 4-week study period.

Anthropometric and body composition measurements including height and weight, waist circumference, bioelectrical impedance will be collected by researcher. Physical activity will be assessed using accelerometers.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-70 yrs BMI 25-39.9kg/m2, Able to attend university for measurement and educational sessions.

Exclusion Criteria:

Cardiovascular problems or documented history of CVD including: angina; myocardial infarction; coronary revascularization procedures; stroke (ischemic or haemorrhagic, including transient ischemic attacks) symptomatic peripheral artery disease that required surgery or was diagnosed with vascular imaging techniques; ventricular arrhythmia; uncontrolled atrial fibrillation; congestive heart failure; hypertrophic myocardiopathy, or aortic aneurism,

Active malignant cancer or history of malignancy within the last 5 years (except non-melanoma skin cancer)

Issues affecting food intake e.g. dysphagia, severe allergies, food neophobia, strong dislike of foods in diet plan, or religious issues

Lack of motivation to change diet/lifestyle (low likelihood as calculated according to the Prochaska and DiClemente Stages of Change Model)

Lack of motivation to fast Medical reasons not allowing very low calorie intake, type 1 or 2 diabetes

Pregnancy or hoping to become pregnant, or breastfeeding

Current adherence to other weight loss or exercise program

Illiteracy or inability/unwillingness to give written informed consent or communicate with study staff

Institutionalization

History of surgical procedures for weight loss or intention to undergo bariatric surgery in the next 12 months

Obesity of known endocrine origin (e.g. hypothyroidism, polycystic ovarian syndrome)

Serious psychiatric disorders including: schizophrenia, bipolar disorder, eating disorders, or depression with hospitalization within the last 6 months

Alcohol abuse or addiction (or total daily alcohol intake >50 g) or drug abuse within the past 6 months

Current use of weight loss medication

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of intervention | 4 weeks
  Participants will complete a questionnaire directed to obtain early markers of how the intervention is used

SECONDARY OUTCOMES:
Total cholesterol | 4 weeks
  Plasma levels of total cholesterol
Weight change | 4 weeks
  Weight change after intervention
Change from baseline dietary intake | 4 weeks
  Participants will self-report dietary intake using the 24-hour dietary recall method. Three days (including 2 weekdays and 1 weekend day) of dietary intake at baseline and after two months will be reported.
Change from baseline physical activity levels at 2 months | 4 weeks
  Physical activity will be assessed assessed during seven days at baseline and after 2 months interventions by accelerometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Applied Sciences, Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No